CLINICAL TRIAL: NCT00527280
Title: Face Reconstruction by Allotransplantation of Composite Tissues
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P050303
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Reconstruction of the Face
Keywords: Allotransplantation:composite tissue; Face transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Feasibility ot face transplantation

INTERVENTIONS:
Procedure: Feasibility ot face transplantation — Feasibility ot face transplantation

SUMMARY:
To show the feasibility of face transplantation in patients

DETAILED DESCRIPTION:
Most facial defects can be reconstructed with autologous tissues using standard plastic surgical techniques. However, when the circular facial muscles (eg. orbicularis oculi and orbicularis oris) are destroyed by burns, ballistic traumas, tumors, or congenital deformities there are no conventional surgical solutions. The study was designed following the advice of the French National Ethics Advisory Committee for life sciences and health (CCNE). The objectives are to study the feasibility and efficacy of face CTA transplantation, functional results, and influence on quality-of-life, as well as the management of immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 65 years
* Signed written informed consent
* patient with a loss of substance of the median third of the face by traumatisms or not carrying the totality of the lips with or without the nasal pyramid.
* validation of the feasibility by a committee of expert in plastic surgery and maxillofacial
* patient with a positive psychologic evaluation
* patient with an anatomical evaluation and assessment pretransplantation positive normal infectious assessment
* Good compliance and capacity of adaptation to the assessment difficulties
* Patient with renal, hepatic, hematologic ,cardiac normal
* Patient profiting from a Social Security cover
* Patient informed patient, having signed a free assent lit with inclusion in the study

Exclusion Criteria:

* patient minor under supervision or deprived of freedom by court order or administrative.
* person remaining in a medical or social establishment
* pregnant. or breast-feeding women
* patient presenting a sever cardiac pathology having a risk of decompensation into pre, per and post operational
* patient presenting a hepatic pathology
* Any cancer that has been in complete remission for > 5 years malignancies tumoral lesion of the face with 2 years deadline of remission respected renal insufficiency chronic clearance of creatin < 60l ml/mn
* chronic respiratory insufficiency
* patient presenting an active infection which can be worsened by the immunosuppression
* patient presenting an active infection which can be worsened by the corticoid
* patient with affection being able to compromise post-operative survival
* patient with digestive ulcer
* No known HIV infection
* serology hepatitis B with circulating DNA highlighted quantitatively
* personality emotional unstable
* schizophrenic or not schizophrenic psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reconstruction tissular at carrier patients of a loss of substance of the median third(third party) of the face having taken the totality of lips with or without the nasal pyramid; or of a loss of substance taking the totality of 4 eyelids. | during the study

SECONDARY OUTCOMES:
To evaluate the potential benefit of such a transplantation in term of quality of life | during the study
To measure the impact of this improvement | during the study
To measure the impact of a immunosuppressive treatment for a pathology which is not vital | during the study
To evaluate Acute Graft rejection using skin and mucosa biopsies: function of the lips and or eyelids mobility and function of the orbicularis muscles Quality of life the psychiatric and psychological evaluations | at in the following days weeks and month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laurent LANTIERI, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital européen Geroges Pompidou, Paris, France

REFERENCES:
- [Derived] Lantieri L, Grimbert P, Ortonne N, Suberbielle C, Bories D, Gil-Vernet S, Lemogne C, Bellivier F, Lefaucheur JP, Schaffer N, Martin F, Meningaud JP, Wolkenstein P, Hivelin M. Face transplant: long-term follow-up and results of a prospective open study. Lancet. 2016 Oct 1;388(10052):1398-1407. doi: 10.1016/S0140-6736(16)31138-2. Epub 2016 Aug 25. PMID 27567680